CLINICAL TRIAL: NCT00903032
Title: Patient-Centered Adherence Intervention After ACS Hospitalization
Brief Title: Patient-Centered Adherence Intervention After Acute Coronary Syndrome (ACS) Hospitalization
Acronym: MEDICATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 08-302
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-09

CONDITIONS: Acute Coronary Syndrome
Keywords: compliance/adherence
MeSH Terms: conditions — Acute Coronary Syndrome; Patient Compliance | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
  Interventions: Behavioral: Intervention
- Arm 2 (Active Comparator): Patients will receive usual care following ACS hospital discharge
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Intervention — The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
  Arms: Arm 1
Behavioral: Usual care — Usual care following ACS hospital discharge.
  Arms: Arm 2

SUMMARY:
We propose to test the effectiveness of a multi-faceted patient-centered adherence intervention among veterans following ACS hospitalization to improve adherence to cardioprotective medications (primary aim). Secondary aims will assess whether the intervention improves achievement of secondary prevention blood pressure (BP) and low density lipoprotein (LDL)-cholesterol goals, reduces cardiac endpoints (myocardial infarction ) MI hospitalization, coronary revascularization, all-cause mortality) and is cost-effective.

ANTICIPATED IMPACT(S) : If successful, the proposed intervention will increase adherence to cardioprotective medications (i.e., -blockers, statins, clopidogrel, and ACE inhibitors) by helping veterans take their medications routinely as prescribed, the quality of cardiovascular care for veterans by helping patients achieve BP and LDL goals which have been associated with improved outcomes, and the efficiency of care by using telephone calls and tele-monitoring for communication with patients rather than clinic visits. The findings of the study will address an important gap in knowledge (i.e., how to improve adherence to medications following ACS discharge) and will be generalizable to other VA Medical Centers and veterans.

DETAILED DESCRIPTION:
RATIONALE: Acute coronary syndrome, including acute myocardial infarction (MI) is one of the leading causes of hospitalization for veterans. Recent advances in the treatment of acute MI have led to declines in hospital mortality. Despite this, the risk of recurrent events and mortality after the index MI hospitalization remains substantial in the following year. Non-adherence to proven cardioprotective medications is a potentially modifiable risk factor that contributes to the persistently high risk of adverse outcomes following MI hospitalization. Prior interventions to improve medication adherence in cardiovascular populations have produced mixed results and have not specifically targeted patients after acute coronary syndrome (ACS) hospital discharge. It is currently unknown if interventions targeting medication non-adherence in the year after ACS discharge will improve medication adherence and intermediate outcomes or will be cost-effective

OBJECTIVE(S): We propose to test the effectiveness of a multi-faceted patient-centered adherence intervention among veterans following ACS hospitalization to improve adherence to cardioprotective medications (primary aim). Secondary aims will assess whether the intervention improves achievement of secondary prevention blood pressure (BP) and LDL-cholesterol goals, reduces cardiac endpoints (MI hospitalization, coronary revascularization, all-cause mortality) and is cost-effective.

METHODS: We propose a 3-year, multi-site patient-level randomized controlled trial to evaluate, relative to usual care, a multi-faceted patient-centered intervention to improve adherence to cardioprotective medication among veterans following ACS hospital discharge. The study will enroll 280 patients to intervention versus usual care for 12-months at 3 VA Medical Centers (Eastern Colorado, Pudget Sound, and Central Arkansas). The proposed intervention will be based on several conceptual frameworks (Chronic Care Model and Medication Adherence Model) and adapt elements of prior successfully adherence interventions, including: collaborative care, patient education, tailoring of medication regimens, and tele-monitoring. The primary analyses will be a comparison of adherence to cardioprotective medications using pharmacy refill records based on the ReCOMP adherence measure developed in the VA. Secondary analyses will compare achievement of secondary prevention BP and LDL goals and cardiac events. In addition, cost-effectiveness analysis will be performed. All analyses will be intention to treat

ELIGIBILITY:
Inclusion Criteria:

All patients admitted with acute coronary syndrome (ACS) as the primary reason for hospital admission and use the VA for their usual source of care, defined as having 1 primary care visit within the 12 months prior to hospital admission will be screened for eligibility to participate. ACS is defined as acute myocardial infarction (both ST-elevation MI and non-ST elevation MI) or unstable angina. The presence of acute myocardial infarction will be defined using standard definitions from an international consensus statement, based on the following: a rise and/or fall of cardiac biomarkers (preferably troponin) with at least one value above the 99th percentile of the upper reference limit and at least one of the following:

* symptoms of ischemia;
* ECG change indicative of new ischemia (new ST-T changes or new left bundle branch block);
* development of pathological Q waves in the ECG; or
* imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.42 Unstable angina will be defined by presence of ischemic symptoms and ECG changes indicative of new ischemia but without biomarker evidence of myonecrosis (i.e., biomarker elevation) and no evidence of new pathological Q waves, loss of viable myocardium or regional wall motion abnormality.

Exclusion Criteria:

* Patient admitted for primary non-cardiac diagnosis and develop ACS as a secondary condition (e.g. perioperative MI);
* planned discharge to nursing home or skilled nursing facility;
* irreversible, non-cardiac medical condition (e.g. metastatic cancer) likely to affect 6-month survival or ability to execute study protocol;
* lack of telephone/cell phone;
* VA is not primary source of care;
* regularly fill medications at non-VA pharmacy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ho, MD PhD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (4):
- United States (4):
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Background] Lambert-Kerzner A, Del Giacco EJ, Fahdi IE, Bryson CL, Melnyk SD, Bosworth HB, Davis R, Mun H, Weaver J, Barnett C, Radcliff T, Hubbard A, Bosket KD, Carey E, Virchow A, Mihalko-Corbitt R, Kaufman A, Marchant-Miros K, Ho PM; Multifaceted Intervention to Improve Cardiac Medication Adherence and Secondary Prevention Measures (Medication) Study Investigators. Patient-centered adherence intervention after acute coronary syndrome hospitalization. Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):571-6. doi: 10.1161/CIRCOUTCOMES.111.962290. PMID 22811499
- [Result] Ho PM, Lambert-Kerzner A, Carey EP, Fahdi IE, Bryson CL, Melnyk SD, Bosworth HB, Radcliff T, Davis R, Mun H, Weaver J, Barnett C, Baron A, Del Giacco EJ. Multifaceted intervention to improve medication adherence and secondary prevention measures after acute coronary syndrome hospital discharge: a randomized clinical trial. JAMA Intern Med. 2014 Feb 1;174(2):186-93. doi: 10.1001/jamainternmed.2013.12944. PMID 24247275
- [Result] Valle JA, Ho PM. Medication adherence in secondary prevention post-myocardial infarction. Curr Treat Options Cardiovasc Med. 2014 Dec;16(12):349. doi: 10.1007/s11936-014-0349-7. PMID 25341689

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Centered Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
  Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of re
- Usual Care: Patients will receive usual care following ACS hospital discharge
  Usual care: Usual care following ACS hospital discharge.
Period: Overall Study
Arm/Group | Patient Centered Intervention | Usual Care
Started | 129 | 124
Completed | 122 | 119
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Patient Centered Intervention: The multi-faceted patient centered intervention adapts elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, PCPs, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens, and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs. Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care, patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
- Total: Total of all reporting groups
Arm/Group | Patient Centered Intervention | Usual Care | Total
Number analyzed (Participants) | 122 | 119 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 73 | 150
  >=65 years | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.57) | 63.8 (9.25) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 120 | 116 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 86 | 84 | 170
  Unknown or Not Reported | 33 | 28 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 9 | 12 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 12 | 29
  White | 92 | 78 | 170
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 14 | 18
Region of Enrollment [Number; unit: participants]
  United States | 122 | 119 | 241

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Cardioprotective Medications (Clopidogrel, Statins, Beta Blockers, ACE-inhibitor/ARB)
Description: The primary outcome was the proportion of patients who were adherent to cardioprotective medications (beta-blockers, statins, clopidogrel, and ACE/ARB) in the year following ACS hospitalization.
Time Frame: 12-months
Population: Composite Adherence* (PDC>0.80) (%)
Measure: Number; unit: percentage of participants
Groups:
- Patient Centered Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
  Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care, patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens, and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
Arm/Group | Patient Centered Intervention | Usual Care
Number analyzed (Participants) | 122 | 119
percentage of participants | 89.3 | 73.9
Statistical Analysis 1: Comparison: Patient Centered Intervention vs Usual Care; Unpaired t tests were used to compare continuous variables, and χ2 testswere used to compare categorical variables across the intervention and usual care. We used a log-rank test to compare the hazardof first hospitalization for MI, revascularization, or death.We used a Wilcoxon rank sum test to compare PDCs between study arms. For all other outcomes, χ2 tests and t testswere used for comparisons, as appropriate; Test type: Non-Inferiority or Equivalence — Previously provided; p = 0.003, Chi-squared

ADVERSE EVENTS:
Groups:
- Patient Centered Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care (between pharmacists, primary care providers, and cardiologists), patient education (tailored to patient needs and provided on a regular ongoing basis), tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
  Intervention: The multi-faceted patient centered intervention will adapt elements of prior successfully adherence interventions and include the following core components: collaborative care, patient education, tailoring of medication regimens (i.e., simplification of dosing, use of pill boxes, synchronization of refill dates), and tele-monitoring via IVR technology as well as patient-specific aides based on identified needs.
Arm/Group | Patient Centered Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/119
Other Adverse Events (participants affected / at risk) | 0/122 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes